CLINICAL TRIAL: NCT06969235
Title: Examining the Role of Executive Functioning in Family-Based Intensive Health Behavior and Lifestyle Treatment to Address Pediatric Obesity (Healthy LIFT Groups)
Brief Title: Examining the Role of Executive Functioning in Family-Based Intensive Health Behavior and Lifestyle Treatment
Acronym: Healthy LIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Crystal Lim, Chair and Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2122709
Record Dates: First submitted 2025-04-30; First posted 2025-05-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IHLBT (Experimental): intensive health behavior and lifestlye treatment
  Interventions: Behavioral: intensive health behavior and lifestyle treatment

INTERVENTIONS:
Behavioral: intensive health behavior and lifestyle treatment — the IHLBT will consist of 18 group meetings over 6 months that teens and parents attend. Topics covered during the meetings will include discussions regarding nutrition and physical activity recommendations, family communication, and use of strategies like monitoring, planning, goal setting, and problem solving.

SUMMARY:
The objectives of this open trial feasibility study are to examine the impacts of intensive health behavior and lifestyle treatment (IHBLT) on youth and caregiver executive functioning (EF), weight status, health behaviors (dietary intake, disordered eating, physical activity), and psychological functioning. Investigators propose to enroll 10 youth 13 to 17 years of age who have overweight or obesity (OV/OB) and a primary caregiver. Families will receive six months of evidence-based family focused group IHBLT based on social, cognitive, and family systems theories. Families will complete assessments of EF skills (objective and self-report), weight status, dietary intake, physical activity, and psychological functioning at pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Youth 13-17 years old
* Youth with OV/OB (BMI≥85th percentile for age/gender norms)
* Participating caregiver must be the participating youth's legal guardian
* Participating youth and caregiver speak and read English
* Participating youth and caregiver agree to attend IHBLT group meetings in-between the pre- and post-treatment assessments.

Exclusion Criteria:

* Youth pervasive developmental disorder (e.g., intellectual disability)
* Youth or caregiver in commercial weight loss program or taking prescribed medications for the prior three months that impact appetite or weight
* Youth or caregiver with documented history of eating disorder or untreated severe depression
* Both youth and caregiver scores are two standard deviations or above the mean on the CPT-3 Commissions and Stroop Interference, representing significantly higher than average EF skills.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Youth EF - CPT-3 Commissions | Post-Treatment (Month 6)
  Youth T-score on the Continuous Performance Test Third Edition (CPT-3) Commissions subscale; T-scores (M = 50, SD = 10) used with higher scores representing worse executive functioning (EF)
Youth EF - Stroop | Post-Treatment (Month 6)
  Youth T-score on the Stroop Color Word Interference scale; T-scores (Mean = 50, SD = 10) used, with higher scores indicating better executive functioning (EF)
Youth EF - Trails B | Post-Treatment (Month 6)
  Youth Trails B z-score; z-score (Mean = 0, SD = 1), with lower scores indicating worse executive functioning (EF)
Youth EF - BRIEF-2 Self Report GEC | Post-Treatment (Month 6)
  Youth self-report on the Behavior Rating Inventory of Executive Function Second Edition (BRIEF-2) Global Executive Composite (GEC) subscale T-score; T-score (Mean = 50, SD = 10), with higher scores representing worse executive functioning (EF)
Youth EF - BRIEF-2 Parent Report GEC | Post-Treatment (Month 6)
  Parent-report of youth Global Executive Composite (GEC) subscale T-score on the Behavior Rating Inventory of Executive Function Second Edition (BRIEF-2); T-score (Mean = 50, SD = 10), with higher scores representing worse executive functioning (EF)

SECONDARY OUTCOMES:
Youth Weight Status | Post-Treatment (Month 6)
  Youth body mass index (BMI) BMI z-score calculated based on height and weight measurements; z-scores have Mean = 0 and SD = 1; higher scores indicate higher weight status
Youth Dietary Intake | Post-Treatment (Month 6)
  Youth Total kcals from 24 hour dietary recall
Youth Physical Activity | Post-Treatment (Month 6)
  Youth time spent in moderate/vigorous physical activity on BLOCK screener

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Lim, PhD, ABPP, Principal Investigator — University of Missouri-Columbia
Locations (1):
- College of Health Sciences, University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No